CLINICAL TRIAL: NCT05004090
Title: Emotional-behavioral Regulation in Children With Neurodevelopmental Disabilities: an Exploratory Investigation of the Role of Genomic Variation, Proteomic Patterns, and Quality of Early Experience
Brief Title: Emotional Regulation in Children With ND: the Role of Genomic Variation, Proteomic Patterns, and Early Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: RC2021_820
Record Dates: First submitted 2021-07-30; First posted 2021-08-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Neurodevelopmental Disabilities; Emotional Regulation; Epigenetics; Parental Factors
MeSH Terms: conditions — Emotional Regulation | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with ND: children with neurodevelopmental disabilities (ND) age between 3 and 24 months (chronologically or corrected in the case of children born preterm).
  Interventions: Diagnostic Test: DNA methylation analysis; Diagnostic Test: Proteomics analysis; Diagnostic Test: Still Face Paradigm
- Typical developed children (TD): children with typical development age between 3 and 24 months (chronological).
  Interventions: Diagnostic Test: DNA methylation analysis; Diagnostic Test: Proteomics analysis; Diagnostic Test: Still Face Paradigm

INTERVENTIONS:
Diagnostic Test: DNA methylation analysis — Genomic DNA will be extracted from 0.4 ml aliquots of each saliva sample using the kit manufacturer's suggested protocol, quantified with Qubit 2.0 (Invitrogen), and stored at -20°C. Aliquots of 250 ng of each DNA will be edited for methylation analysis with the EZ DNA Methylation Lightning kit (Zymo Research). Amplification of samples and their preparation for NGS sequencing will be performed as described. Samples will be sequenced on NextSeq 500 (Illumina). Individual processed sequences (PE reads) will be independently aligned to reference sequences using a parallel Smith-Waterman algorithm. Only reads that consistently align to the same reference sequence will be retained. At each CpG site in each analyzed sequence, the frequencies of the four bases will be evaluated and tabulated.
Diagnostic Test: Proteomics analysis — Urine samples are collected using non-invasive methods and are prepared according to a procedure preparatory to quantitative recovery of exosomes: once thawed and centrifuged at 17,000 x g for 10 min at 4°C, the recovered supernatants are separated and centrifuged at 200,000 x g for 1 hr at 4°C. Exosome pellets are separated, washed repeatedly and resuspended in buffer (NH4HCO3, 0.1 mM ph=7.8). Protein concentration is estimated with the SPNTM Protein Assay kit and each sample (50 ± 0.5 μg protein) is digested with trypsin using a 1:50 (w/w) enzyme/substrate ratio at 37 °C over night (o/w). A second tryptic digestion is performed with an enzyme:substrate ratio of 1:100 (w/w) for 4h. Digested samples, centrifuged at 13,000 × g for 10 min, are purified and concentrated using PepClean C-18 columns. The samples obtained are analyzed by reversed-phase liquid chromatography coupled to high-resolution mass spectrometry.
Diagnostic Test: Still Face Paradigm — During an observational session, a short video recording of the mother-child interaction of approximately 10 minutes will be made in a semi-structured setting to assess the child's emotional regulation and social behavior. The interaction will be structured in 5 different phases according to the Still Face paradigm (Tronick et al., 1978): Play, Still#1, Reunion#1, Still#2, Reunion#2. Play: Mothers will be invited to interact with their babies for 10 minutes; Still: mothers will be asked to remain still while maintaining an unresponsive expressionless face and not to smile, touch, or talk to the child for 2 minutes (Still#1: 2 minutes; Still#2: 2 minutes); Reunion: mothers will be asked to resume the play activity with their own for an additional 2 minutes (Reunion#1: 2 minutes; Reunion#2: 2 minutes).

SUMMARY:
Children with neurodevelopmental disabilities (ND) represent an heterogeneous population characterized by a wide range of clinical diagnoses (e.g., cerebral palsy, sensory impairment, psychomotor retardation), which are associated with various deficits that emerge early in the child's life. Although it has been broadly demonstrated that children with ND exhibit several differences in social-emotional skills and emotional-behavioral regulation, the underlying mechanisms that are associated with more or less impaired developmental trajectories remain still partially unexplored. While several studies have investigated the role of biological and environmental factors in the emotional behavioral regulation of typically developing children or children with risk conditions other than ND (e.g., children who are victims of maltreatment), little research has jointly explored the role of methylation, polymorphisms, and environmental experience in the emotional-behavioral regulation of children with ND during the first years of life. The aim of this project is to investigate biological (DNA methylation, polymorphic variants, and proteomics) and environmental (e.g., painful and/or invasive nursing procedures, proximity, and physical contact) factors that might be associated with the emotional behavioral regulation of children with ND.

DETAILED DESCRIPTION:
Background: Children with neurodevelopmental disabilities (ND) are an heterogeneous population characterized by a wide variety of clinical diagnoses, which are associated with different deficits that emerge during infancy and childhood. Although diagnostic framing may vary, several studies observed that children with ND share reduced social-relational skills, characterized by lower interactive and dyadic attention skills and decreased use of interpersonal communication cues. Although it has been broadly demonstrated that children with ND exhibit several differences in social-emotional skills and emotional behavioral regulation, the underlying mechanisms that are associated with more or less impaired trajectories remain partially unexplored.

Primary aim: to explore in a sample of children with ND aged 3 to 24 months the contribution of 1) methylation of candidate genes (e.g., OXTR, SLC6A4, BDNF, and DRD4), 2) polymorphisms in emotional-behavioral regulation, and 3) environmental experience (i.e., adverse experiences and quality of parental behavior) in emotional-behavioral regulation.

Secondary aim: 1) to explore a possible association between proteomics and emotional-behavioral regulation in a sample of children with ND aged between 3 and 24 months; 2) to identify functional and structural patterns of candidate genes associated with emotional behavioral regulation by applying a computational approach. Modules of genes potentially associated with social-emotional development in networks of interaction and spatio-temporal co-expression in the encephalon will also be identified.

Planned Activities:

Methods:the project involves a clinical group of children with ND and their mothers and a control group of typically developing children and their mothers. Because of the nature of the groups, the study is a quasi-experimental research design.

The study involves the following procedures:

* collection of biological material: saliva collection using non-invasive modalities and the Oragene OG575 kit (Genotek DNA) and urine collection using non-invasive modalities.
* administration of questionnaires and diary of proximity: the mother (both for the clinical group and for the control group) will be asked to fill out some questionnaires relating to their mood, habitual behavior and development of the child. It will also be evaluated how much and in what way the mother spends in physical contact (e.g. time spent caressing the baby; time spent holding the baby; time spent when the baby is attached to the mother's breast). This data will be derived through the use of a repurposed version of Raiskila et al.'s "closeness diary" implemented in an electronic format, in the form of an APP (APP: inContatto);
* videotaping the Parent-Child Interaction in a semi-structured context in 5 different phases in accordance with the Still Face paradigm (Tronick et al., 1978): Play, Still#1, Reunion#1, Still#2, Reunion#2.

Interactions will be videotaped for subsequent behavioral coding using various coding tools. The child's emotional-behavioral regulation will be coded using the coding systems: a) Infant and Caregiver Engagement Phase, b) Infant Regulatory Scoring System and Maternal Regulatory Scoring System by Tronik. In addition, infant and maternal behavior will be coded using the Global Rating Scale coding system by Murray and maternal touch behavior using the Maternal Touch Coding System by Provenzi.

ELIGIBILITY:
Inclusion Criteria:

Children with ND:

* Age between 3 and 24 months (chronologically or corrected in the case of children born preterm);
* mild to moderate developmental delay documented by clinical signs (e.g., symptoms of brain injury on neurological examination or neuroimaging) or by developmental scales (i.e., Griffiths III scales) associated with various diagnoses (e.g., cerebral palsy, prematurity);
* absence of genetic syndromes. The Griffiths III scale will be used to assess the child's overall level of development.

Typical developmental children:

* birth to term;
* age between 3 and 24 months (chronological);
* absence of peri- or postnatal pathology.

Inclusion criteria for mothers (DN and typical development):

* age above 18 years;
* good understanding of the Italian language;
* absence of cognitive difficulties and/or psychiatric disorders;
* no intake of psychotropic medications;
* not part of a single-parent family.

Exclusion Criteria: refer to the inclusion criteria.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with ND and their mothers will be recruited through consecutive and convenience sampling at the U.O.C. "Specialistic Rehabilitation - Neuropsychiatric Pathologies of Developmental Age" and the U.O.C. "Functional Rehabilitation" of the Scientific Institute "E. Medea" (Bosisio Parini site). Children with typical development and their mothers will be recruited from nursery schools in the province of Lecco. After viewing an informative letter describing the general research, mothers will be contacted by telephone and invited to participate voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant DNA methylation status | 1 day , at the recruitment
  The DNA methylation status (i.e. percentage) of candidate genes (e.g., OXTR, SLC6A4, BDNF, and DRD4) will be assessed from salivary samples obtained from infants.
Infant behavioral regulation | 1 day , at the recruitment
  The infant behavioral regulation (i.e., negative emotionality) will be coded micro-analitically (i.e., second-by-second) from videotapes of mother-infant interactions.

SECONDARY OUTCOMES:
Infant proteomic patterns | 1 day , at the recruitment
  Proteomic patterns will be evaluated for the relative amount and post-translational modifications of candidate proteins, thought to be involved with the stress response in infants.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy